CLINICAL TRIAL: NCT05126537
Title: An Observational Study on the Relationship Between Expression of Co-inhibitory Molecules on Treg and miR-155-5p Expression in the Peripheral Blood of Patients With Sepsis
Brief Title: Co-inhibitory Molecules on Treg and miR-155-5p in Patients With Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Songqiao Liu, Chief, Southeast University, China
Other Study IDs: 2020ZDSYLL041-Y01
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: 28 Day Mortality
Keywords: sepsis immunosuppression Treg

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — Venous blood was extracted according to time points and stored
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Health volunteers: Health volunteers as control group
  Interventions: Other: no intervention
- ICU non-sepsis patients: ICU non-sepsis patients as control group
  Interventions: Other: no intervention
- Sepsis patients: Sepsis patients as study group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — prospective and observational study with no intervention

SUMMARY:
there is high mortality rate of sepsis, 36% in 90-days of sepsis in China, and there is no effective treatment. Immunosuppression mediated by sepsis is an important cause of death in patients. Treg cells are important immunomodulatory cell. Treg's over-differentiation is involved in the development of sepsis induced immunosuppression. In sepsis patients, the expression of PD-1、CTLA-4 and TIGIT on Treg cell surface increased, and Treg cells with high expression of co-inhibitory molecules showed stronger immunosuppressive characteristics. MiR-155-5p is an unencoded RNA transcript from a proto-oncogene B cell integration cluster. In sepsis, the expression of miR-155 increased in peripheral blood and correlated with the patient's prognosis. Recent studies have shown that miR-155-5p promotes co-inhibitory molecules expressed on T cells in LCMV infected animal models. However, the relationship between the expression of peripheral blood miR-155-5p in sepsis patients and the expression of co-inhibitory molecules on Treg cell surface is not clear.

DETAILED DESCRIPTION:
1. peripheral blood Treg cells and their surface PD-1、CTLA-4 and TIGIT levels in sepsis patients were measured by flowcytometry. SOFA score、APACHE II score were recorded
2. the level of miR-155-5p were measured by RT-qPCR in patients with sepsis on day 0-1 and day 3-5, and the correlation between the expression of the co-inhibitory molecules and miR-155-5p were evaluated

ELIGIBILITY:
Inclusion Criteria:

* sepsis 3.0 diagnositic criteria are met. older than 18 years old. total course is less than 7 days. Informed consent is obatained.

Exclusion Criteria:

* pregnancy. patients with active malignant tumors. chronic hepatitis or HIV. patients under treatment with immunosuppressive drugs (except patients with glucocorticosteroid prednisone or equivalent dose<10 mg/d per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with sepsis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
28 day mortality | 28 days
  all patients followed up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Qingxiang Liu, MD., Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided